CLINICAL TRIAL: NCT06818318
Title: The Effect of Smartphone Addiction on Temporomandibular Dysfunction
Brief Title: Smartphone Addiction and Temporomandibular Dysfunction
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hazel Çelik Güzel, Assist. Prof. Dr, Bandırma Onyedi Eylül University
Other Study IDs: 2024-27
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Smartphone Addiction
Keywords: smartphone addiction; temporpmandibular disorders; head posture; pain
MeSH Terms: conditions — Internet Addiction Disorder; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Temporomandibular disorder — Fonseca's Anamnestic Index was used for TMJ dysfunction. The diagnostic accuracy of the Fonseca's Anamnestic Index was found to be high in identifying pain-related and intra-articular TMDs, and the cut-off point was set as 25 points. A score of 25 and above was accepted as the presence of TMD.
Other: Smartphone Addiction Scale-Short Form — In our study, the Smartphone Addiction Scale-Short Form will be filled out in order to evaluate the intensity of smartphone use of students, and the daily duration of smartphone use will be recorded. The Smartphone Addiction Scale-Short Form is a 6-point Likert-type scale consisting of 10 items used to measure the risk of smartphone addiction. Scores obtained from the scale vary between 10-60, and an increase in the score indicates an increased risk for smartphone addiction. Although the scale does not have a cut-off score in our country, it was determined as 31 for men and 33 for women in the Korean sample.
Other: Neck Disability Index — The Neck Disability Index was used to assess the disability caused by neck pain. This questionnaire consists of ten items, four of which are related to subjective symptoms (pain intensity, headache, concentration, sleep) and six of which are related to activities of daily living (self-care, lifting, reading, work, driving and leisure activities). Scale scoring ranges from 0-40.
Other: Temporomandibular Joint Pain — Numeric Pain Scale is a simple, reliable and short-term method commonly used in the clinic to measure pain intensity. It is a very reliable method in the evaluation of pharmacological and nonpharmacological treatments that reduce pain. The patient is told that the most severe pain he/she experiences is 10, and if he/she has no pain, the pain intensity is 0. The participant was asked to say a number between 0 and 10 corresponding to the intensity of pain felt in the TMJ region.
Other: Anterior posture of the head — The anterior posture of the head was assessed with the Craniovertebral angle using a goniometer. The Craniovertebral angle was measured in degrees as the angle between the horizontal plane and the 7th cervical vertebra and the ear hole.
Other: Pressure Pain Threshold Assessment — In our study, the pressure pain threshold measurement of the dominant and non-dominant side masseter and tenar muscles was evaluated with Baseline manual algometer.

SUMMARY:
The aim of this study was to investigate the effect of smartphone addiction on temporomandibular dysfunction with the determinants of pain threshold, head posture and neck disability level.

DETAILED DESCRIPTION:
Firstly, the purpose of the research and the evaluation methods were explained to the students. Students who volunteered to participate in the study and met the inclusion criteria were included in the evaluation. Approval was obtained from the evaluated students with the 'Informed Voluntary Consent Form'. Then, the students will fill in the Descriptive Data Form. The risk of smartphone addiction of the students who filled out the Descriptive Data Form was assessed with the Smartphone Addiction Scale-Short Form, TMD dysfunction status was assessed with the Fonseca Anamnestic Index, neck disability status was assessed with the Neck Disability Index, TMJ pain was assessed with the Numeric Pain Scale, head posture was assessed with a goniometer, and pressure pain threshold of the tenar and masseter muscles was assessed with an algometer. The evaluations took an average of 45 minutes for each student. The evaluations of the students were performed only once.

ELIGIBILITY:
Inclusion Criteria:

* To study at Bandirma Onyedi Eylül University
* Students between the ages of 18-30 years, whose voluntary consent was obtained and who use smartphones

Exclusion Criteria:

* Individuals undergoing masseter botox application
* Individuals diagnosed with TMJ disorder and/or bruxism
* Individuals with musculoskeletal system problems such as fractures of the hand, fingers, upper extremities and/or TMJ, rheumatoid disease with evidence of systemic, specific pathological conditions
* Individuals who have undergone any surgical operation related to hand, finger, upper extremity and/or TMJ problem
* Individuals who have received hand, finger, upper extremity and/or TMJ-related physiotherapy and rehabilitation services in less than 6 months
* Individuals with facial paralysis
* Individuals with diagnosed psychiatric illness.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University students
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Temporomandibular disorder | June 1, 2024- December 1, 2024
  Fonseca's Anamnestic Questionnaire was used for TMJ dysfunction. The diagnostic accuracy of the Fonseca's Anamnestic Questionnaire was found to be high in identifying pain-related and intra-articular TMDs, and the cut-off point was set as 25 points. A score of 25 and above was accepted as the presence of TMD.
Smartphone Addiction Scale-Short Form | June 1, 2024- December 1, 2024
  In our study, the Smartphone Addiction Scale-Short Form will be filled out in order to evaluate the intensity of smartphone use of students, and the daily duration of smartphone use will be recorded. The Smartphone Addiction Scale-Short Form is a 6-point Likert-type scale consisting of 10 items used to measure the risk of smartphone addiction. Scores obtained from the scale vary between 10-60, and an increase in the score indicates an increased risk for smartphone addiction. Although the scale does not have a cut-off score in our country, it was determined as 31 for men and 33 for women in the Korean sample.
The Neck Disability Index | June 1, 2024- December 1, 2024
  The Neck Disability Index was used to assess the disability caused by neck pain. This questionnaire consists of ten items, four of which are related to subjective symptoms (pain intensity, headache, concentration, sleep) and six of which are related to activities of daily living (self-care, lifting, reading, work, driving and leisure activities). Scale scoring ranges from 0-40.
Temporomandibular Joint Pain | June 1, 2024- December 1, 2024
  Numeric Pain Scale is a simple, reliable and short-term method commonly used in the clinic to measure pain intensity. It is a very reliable method in the evaluation of pharmacological and nonpharmacological treatments that reduce pain. The patient is told that the most severe pain he/she experiences is 10, and if he/she has no pain, the pain intensity is 0. The participant was asked to say a number between 0 and 10 corresponding to the intensity of pain felt in the TMJ region.
Anterior head posture | June 1, 2024- December 1, 2024
  The anterior posture of the head was assessed with the Craniovertebral angle using a goniometer. The Craniovertebral angle was measured in degrees as the angle between the horizontal plane and the 7th cervical vertebra and the ear hole.
Pressure pain threshold assessment | June 1, 2024- December 1, 2024
  In our study, the pressure pain threshold measurement of the dominant and non-dominant side masseter and tenar muscles was evaluated with Baseline manual algometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Balıkesir, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided